CLINICAL TRIAL: NCT03433014
Title: A Prospective Randomized Controlled Trial of Postoperative Analgesic Effects of Local Wound Infiltration With 0.5% Levobupivacaine in Laparoscopic Colorectal Surgery.
Brief Title: Local Wound Infiltration With 0.5% Levobupivacaine for Postoperative Pain After Laparoscopic Colorectal Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Ramathibodi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016/200
Record Dates: First submitted 2018-01-31; First posted 2018-02-14 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Laparoscopic Colorectal Surgery; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Levobupivacaine

STUDY DESIGN:
Intervention Model Description: The infiltration group will receive local infiltration with 0.5% Levobupivacaine. The trocar insertion sites are infiltrated before the skin incision is made. Using the Lap-Assist Transversus Abdominis Plane Block Technique, the total volume of infiltrated 0.5% Levobupivacaine is 20 ml, divided proportionally according to the length of the skin incision (2 ml for the 5-mm trocar and 3 ml for the 10-mm trocars, and 10 mL for specimen retrieval incision). The control group will not receive any local infiltrative agent.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.5% Levobupivacaine (Active Comparator): The trocar insertion sites are infiltrated before the skin incision is made. Using the Lap-Assist Transversus Abdominis Plane Block Technique, the total volume of infiltrated 0.5% Levobupivacaine is 20 ml, divided proportionally according to the length of the skin incision.
  Interventions: Procedure: 0.5% Levobupivacaine
- Control (Other): The control group will not receive any local infiltrative agent.
  Interventions: Other: Control

INTERVENTIONS:
Procedure: 0.5% Levobupivacaine — The infiltration group will receive local infiltration with 0.5% Levobupivacaine. The trocar insertion sites are infiltrated before the skin incision is made. Using the Lap-Assist Transversus Abdominis Plane Block Technique, the total volume of infiltrated 0.5% Levobupivacaine is 20 ml, divided proportionally according to the length of the skin incision (2 ml for the 5-mm trocar and 3 ml for the 10-mm trocars, and 10 mL for specimen retrieval incision). The specimen retrieval incision will be performed in one of two techniques, depending on the surgeon's preference, a 4-6 cm length midline incision (extending from the Hasson trocar incision) or a 4-6 cm length Pfanensteil incision.
  Arms: 0.5% Levobupivacaine
Other: Control — No infiltration
  Arms: Control

SUMMARY:
The study design is a prospective randomized, double-blind, controlled trial of patients who are due to have elective laparoscopic colorectal surgery in Ramathibodhi Hospital. The primary objective is to measure pain scores (Visual Analog Scale) in the postoperative period. The secondary objective is to compare the VAS scores between the two types of technique used for specimen retrieval incision.After approval by the ethics committee, patients scheduled for elective laparoscopic colorectal surgery under general anesthesia who are eligible for inclusion criteria were recruited for this study after informed consent by surgical residents or surgical staff at the Outpatient Department (OPD). Patients who meet the exclusion criteria will be excluded.

DETAILED DESCRIPTION:
During a preoperative visit, the patients are introduced to the concept of the visual analogue scale (VAS), which ranges from 0 = no pain to 10 = worst pain.

Once given general anesthesia in the operating room, the patient will be randomly selected into one of the two arms of this report's diagram (1:1 ratio) through the drawing of a sealed, opaque envelope by one of the surgical residents in charge or by the attending surgeon. The infiltration group will receive local infiltration with 0.5% Levobupivacaine. The trocar insertion sites are infiltrated before the skin incision is made. Using the Lap-Assist Transversus Abdominis Plane Block Technique, the total volume of infiltrated 0.5% Levobupivacaine is 20 ml, divided proportionally according to the length of the skin incision (2 ml for the 5-mm trocar and 3 ml for the 10-mm trocars, and 10 mL for specimen retrieval incision). The control group will not receive any local infiltrative agent.After induction, the pneumoperitoneum will be created via the Open Hasson Technique and using a 10-12-mm trocar. During surgery, intraabdominal pressure is maintained at 12-15 mmHg. In addition to the Hasson trocar, one 10-mm and two to three 5-mm trocars will be used. The specimen retrieval incision will be performed in one of two techniques, depending on the surgeon's preference, a 4-6 cm length midline incision (extending from the Hasson trocar incision) or a 4-6 cm length Pfanensteil incision.

A standardized plan for postoperative analgesia is prepared. All patients will receive one 500 mg tablet of oral paracetamol every 6 hours when postoperative oral intake is allowed by the attending doctor. In patients with VAS scores >3, parenteral opioid (Morphine) is given.

The hospital volunteer nurses caring for the patients during the preoperative and postoperative course are given standard pain evaluation protocols. All study pain evaluators and patients are blinded to treatment assignments throughout the pain assessment process.

After the operation, the inpatient ward nurse will record the patients' pain score at 4 hours after surgery using the VAS score and record the results in the study data recording form attached to each patient's medical record chart. Additional morphine usage data is also recorded.

All side effects, such as tinnitus, nausea, vomiting, headache, dizziness, seizure, cardiovascular instability, and local wound complication will be recorded and treated by the attending resident or consultant doctor.

All data is collected by the main investigator from the patient chart and data recording form. Data is expressed as mean ± SD. Parametric data is compared between groups. Statistical significance is set at a level of p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic colorectal surgery under general anesthesia.
* ASA (American Society of Anesthesiologists) classification 1 and 2
* Laparoscopic colorectal surgery including Laparoscopic segmental colonic resection, laparoscopic anterior resection and laparoscopic low anterior resection

Exclusion Criteria:

* Conversion to open surgery.
* Patients receive epidural anesthesia.
* Patients have history allergy to aminoamides.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-31 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
measure pain scores (Visual Analog Scale) in the postoperative period | 4 hours after surgery using the VAS score
  After the operation, the inpatient ward nurse will record the patients' pain score at 4 hours after surgery using the VAS score and record the results in the study data recording form attached to each patient's medical record chart.standardized plan for postoperative analgesia is prepared. All patients will receive one 500 mg tablet of oral paracetamol every 6 hours when postoperative oral intake is allowed by the attending doctor. In patients with VAS scores >3, parenteral opioid (Morphine) is given.

SECONDARY OUTCOMES:
objective is to compare the VAS scores between the two types of technique used for specimen retrieval incision | 4 hours after surgery using the VAS score
  The secondary objective is to compare the VAS scores between the two types of technique used for specimen retrieval incision.. The specimen retrieval incision will be performed in one of two techniques, depending on the surgeon's preference, a 4-6 cm length midline incision (extending from the Hasson trocar incision) or a 4-6 cm length Pfanensteil incision.

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Supsamutchai, MD, Study Chair — Ramathibodi Hospital, Mahidol University; Chumpon Wilasrusmee, MD, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Chairat Supsamutchai, Bangkok, Bankok, Thailand

IPD SHARING:
Plan to Share IPD: No